CLINICAL TRIAL: NCT04535414
Title: Phase II Randomized Trial of Bethesda Protocol Compared to Cambridge Method for Detection of Early Stage Gastric Cancer in CDH1 Mutation Carriers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Blakely, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 200150; 20-C-0150
Record Dates: First submitted 2020-09-01; First posted 2020-09-02 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer; Gastric Neoplasms; Gastric Adenocarcinoma
Keywords: Diagnostic; Diagnosis; HDGC; SRCC; Confocal Endoscopic Microscopy (CEM)
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1/ Arm 1: Bethesda Protocol (investigational) with Confocal Endomicroscopy (Experimental): Bethesda protocol (investigational) with confocal endomicroscopy in assigned participants
  Interventions: Device: Cellvizio (Registered trademark) Real-Time In Vivo Cellular Imaging Platform with Confocal Miniprobes; Device: Olympus Graphics Interchange Format (GIF) 190 endoscope; Procedure: Gastric mucosal biopsy
- 2/ Arm 2: Cambridge Method (control) with Confocal Endomicroscopy (Active Comparator): Cambridge method (control) with confocal endomicroscopy in assigned participants
  Interventions: Device: Cellvizio (Registered trademark) Real-Time In Vivo Cellular Imaging Platform with Confocal Miniprobes; Device: Olympus Graphics Interchange Format (GIF) 190 endoscope; Procedure: Gastric mucosal biopsy

INTERVENTIONS:
Device: Cellvizio (Registered trademark) Real-Time In Vivo Cellular Imaging Platform with Confocal Miniprobes — Participants of both study arms will undergo confocal endomicroscopy of the gastric mucosa until sufficient data for statistically accurate and reliable application of machine learning (i.e., computer models), currently believed to total the first 50 enrolled participants.
Device: Olympus Graphics Interchange Format (GIF) 190 endoscope — Participants will undergo white light endoscopy. The mucosa of the stomach may be thoroughly washed before examination, as medically indicated, and inspection will include repeated inflation and deflation to check distensibility and any abnormal appearing areas will additionally be biopsied. Nontargeted biopsies will be obtained as indicated per the assigned Arm.
Procedure: Gastric mucosal biopsy — As clinically indicated.

SUMMARY:
Background:

Some people have a mutation in the cadherin-1 gene (CDH1) gene that is known to lead to stomach cancer. They are advised to get regular endoscopies with biopsies even if their stomach appears normal. The endoscopy method currently used is called the 'Cambridge Method.' Researchers want to test a new method called the 'Bethesda Protocol.'

Objective:

To compare the Cambridge Method and Bethesda Protocol and find out which is more efficient in catching early signs of cancer.

Eligibility:

Adults age 18 and older who have a mutation in the CDH1 gene.

Design:

Participants will be screened with a review of their medical history, medical records, and physical status.

Participants will be put into group 1 (Bethesda Protocol) or group 2 (Cambridge Method).

Participants will have a physical exam. They will have endoscopy. For this, they will be put under general anesthesia. They will wear compression cuffs around their legs to prevent blood clots. A lighted tube will be inserted into their mouth and go down to their stomach.

For group 1 participants, 88 pieces of tissue will be taken from 22 areas of their stomach.

For group 2 participants, 30 pieces of tissue will be taken from 6 areas of their stomach. Then group 2 will be injected with a contrast dye. A microscope will be inserted, and more samples will be taken.

About 14 days later, participants will have a follow-up visit or phone call. They may give stool samples every 3 to 6 months for 12 months for research purposes.

Participants may have another endoscopy 6-18 months later.

DETAILED DESCRIPTION:
Background:

Hereditary Diffuse Gastric Cancer (HDGC) is most often attributed to inactivating germline mutations in the E-cadherin (CDH1) tumor suppressor gene. Mutation carriers have a 24-70% lifetime risk of developing gastric adenocarcinoma.

International consensus guidelines recommend endoscopic screening and surveillance of CDH1 mutation carriers who decline risk-reducing total gastrectomy (TG). However, this approach lacks sufficient sensitivity for detection of occult, intramucosal foci of signet ring cancer cells (SRCC), which are pathognomonic of HDGC. Our team has established a systematic endoscopic screening protocol (Bethesda protocol) that demonstrates a higher rate of SRCC detection compared to historic controls using the currently recommended Cambridge method.

Objective:

Determine if Bethesda protocol provides improved sensitivity for detection of early-stage gastric cancer in CDH1 germline mutation carriers compared to the Cambridge method.

Eligibility:

Subjects with pathogenic or likely pathogenic CDH1 germline mutation.

Age >=18 years.

Physiologically able to undergo upper endoscopy

Design:

Phase II randomized study to compare Bethesda protocol and Cambridge method for detection of intramucosal SRCC in asymptomatic CDH1 mutation carriers undergoing endoscopic screening or surveillance.

ELIGIBILITY:
* INCLUSION CRITERIA:
* An individual who harbors a pathogenic, or likely pathogenic, cadherin-1 gene (CDH1) germline variant.

Note: individuals with CDH1 variant classified as any of the following are not eligible:

* variant of uncertain significance
* benign
* likely benign.

  * Age greater than or equal to 18 years.
  * Physiologically able to undergo upper endoscopy.
  * Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Any clinical contraindication (e.g., known bleeding disorder, thrombocytopenia) to endoscopic biopsy.
* Unstable angina or recent (within 3 months) myocardial infarction.
* Any clinical contraindication to general anesthesia.

Re-Enrollment:

INCLUSION CRITERIA:

* Subject must have previously been enrolled on the study and must have undergone endoscopy. Note: Subject may re-enroll only once after initial endoscopy performed
* Subject must have clinical need for a repeat endoscopy
* Prior on-protocol endoscopy must have occurred at least 6 months (+/- 2 weeks) and no greater than 18 months (+/- 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, bacterial gene sequences will be deposited in GenBank.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Bacterial gene sequences data are available once bacterial gene sequences data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Bacterial gene sequences data are made available via GenBank; NCBI places no restrictions on the use or distribution of the GenBank data.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0150.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
Started | 98 | 97
Completed | 89 | 91
Not Completed | 9 | 6
Not completed — Taken off study due to principal investigator (PI) discretion. | 1 | 0
Not completed — Cancelled appointment | 1 | 0
Not completed — cancelled - food in stomach | 2 | 0
Not completed — Study closed per PI decision prior to scheduled intervention | 5 | 5
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 80 | 165
  >=65 years | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.46 (15.89) | 49.84 (13.6) | 47.13 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 42 | 44 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 91 | 92 | 183
  Ethnicity: Unknown or Not Reported | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 88 | 90 | 178
  More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 3 | 0 | 3
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 98 | 97 | 195

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Improved Sensitivity for Detection of Early-stage Gastric Cancer in CDH1 Germline Mutation Carriers Compared to the Cambridge Method
Description: Among participants who undergo gastrectomy, in each of the two arms, the fraction of participants who had signet ring cell carcinoma (SRCCs) previously identified by endoscopic biopsy out of those who had SRCCs detected on final pathologic analysis of gastrectomy explants will be used to determine the difference between 30% sensitivity in the Cambridge method and 60% sensitivity in the Bethesda protocol of each arm on a Fisher's exact test with a 0.05 two-sided significance level and reported with a 95% confidence interval.
Time Frame: 14 days
Population: No participants underwent total gastrectomy in Arm 2.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
Number analyzed (Participants) | 2 | 0
proportion of participants | 1 [0 to 1] |

2. Secondary Outcome: Proportion of Participants Who Had Signet Ring Cell Carcinoma (SRCC) Identified on Final Pathology But Were Negative for SRCC on Esophagogastroduodenoscopy (EGD)
Description: False negative rate of SRCC detection in participants who undergo risk-reducing total gastrectomy using the Bethesda protocol and Cambridge method. The differences in fractions will be compared using a two-tailed Fisher's exact test and reported with a 95% confidence interval.
Time Frame: 14 days
Population: No participants underwent total gastrectomy in Arm 2.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
Number analyzed (Participants) | 2 | 0
proportion of participants | 0.5 [0 to 1] |

3. Secondary Outcome: Difference in Fractions of Participants Crude Cancer Detection Rates Between Endoscopy Using the Bethesda Protocol and the Cambridge Method
Description: The difference in fractions of participants with signet ring cell carcinoma (SRCCs) crude cancer detection rates found on endoscopy by the Bethesda protocol and the Cambridge method determined by the power to detect a difference with a two-sided 0.05 significance level between 15% and 30% crude cancer detection rates and reported with a 95% confidence interval.
Time Frame: 14 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
Number analyzed (Participants) | 89 | 91
proportion of participants | 0.31 [0.24 to 0.46] | 0.20 [0.13 to 0.31]

4. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: From the start of endoscopy through 14 days following study interventions, an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
Number analyzed (Participants) | 98 | 97
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: From the start of endoscopy through 14 days following study interventions, an average of 2 weeks.
Arm/Group | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/97
Other Adverse Events (participants affected / at risk) | 4/98 | 0/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/ Arm 1: Bethesda Protocol (Investigational) With Confocal Endomicroscopy (N=98) | 2/ Arm 2: Cambridge Method (Control) With Confocal Endomicroscopy (N=97)
Fever (General disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04535414/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04535414/ICF_001.pdf